CLINICAL TRIAL: NCT05601453
Title: Evaluation of Clinical Outcomes of Patients Undergoing a Redo-TAVI Procedure; a Multicenter Prospective Observational Registry
Brief Title: The ReTAVI Prospective Observational Registry
Status: Recruiting | Type: Observational
Sponsor: Institut für Pharmakologie und Präventive Medizin (Network)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: ReTAVI Registry
Record Dates: First submitted 2022-10-07; First posted 2022-11-01 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Structural Valve Deterioration; Structural Valve Degeneration; Symptomatic Patients Who Have Had Transcatheter Heart Valve (THV) Failure; Prosthetic Valve Malfunction; Prosthesis Failure
Keywords: Transcatheter Aortic Valve Implantation (TAVI); Structural Valve Deterioration; redo-TAVI; THV-in-THV; TAV-in-TAV; TAVR-in-TAVR; Redo-TAVR; Revalve
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- redo-TAVI patients: Patients with severe aortic stenosis (sAS) treated with TAVI developing SVD and thus an indication for redo-TAVI procedure
  Interventions: Procedure: Elective redo transcatheter aortic valve implantation (redo-TAVI)

INTERVENTIONS:
Procedure: Elective redo transcatheter aortic valve implantation (redo-TAVI) — Elective redo-TAVI procedure with the intention to treat the patient with a SAPIEN family valve implantation (currently the only registered medical devices for redo-TAVI use)
  Other Names: redo-TAVI; redo-TAVR; Valve-in-Valve (ViV); TAV-in-TAV; TAVR-in-TAVR; Revalve

SUMMARY:
Patients with severe aortic stenosis (sAS) treated with transcatheter aortic valve implantation (TAVI) (increasingly younger & lower risk pts) are experiencing SVD of the index THV and thus developing an indication for a redo-TAVI procedure.

The evidence on redo-TAVI (where a transcatheter heart valve [THV] is implanted into another THV) is limited, with initial data showing acceptable safety as well efficacy in highly selected and limited populations.

Aim is to evaluate short- and long-term data on patients undergoing transcatheter redo-TAVI procedures with THVs for failure of a previously implanted THV and to determine VARC-3 defined efficacy and safety at 30 days and functional outcome at 1 year, 3 years and 5 years.

DETAILED DESCRIPTION:
Between 1.4 and 2.8% of all patients undergoing transcatheter heart valve (THV) implantation require a second THV implanted into the previously implanted THV because of clinically significant aortic regurgitation [1-3]. 90% of THV-in-THV implants were considered successful although the mortality in the redo-TAVI group was higher at similar STS risks as in those with a successful first implant.

Redo-TAVI may also be a promising treatment strategy in degenerated THVs, but there is insufficient knowledge which strategy and valve design may result in the best outcomes [4]. Evidence so far reported is based on case reports and small case series, but not on a prospective, multicenter documentation.

Currently, ~ 5% of THV are implanted in degenerated surgical bioprosthetic valves. With the expanded use of THV for treatment of lower risk patients with severe aortic stenosis (sAS), it is estimated that the number of patients requiring re-treatment for THV failure is likely to rise within the next years.

ELIGIBILITY:
Inclusion Criteria:

Consecutive patients fulfilling the following criteria:

1. Consenting adult patient (≥18 years)
2. Procedural success of the first TAVI
3. TAVI device failure of the index THV, irrespective of SVD severity
4. Intention to treat the patient with a redo-TAVI procedure (SAPIEN family THV)
5. The Local Heart Team and the Case Review Board consider the patient suitable and indicated for elective redo-TAVI
6. Patient is scheduled to undergo a 30 Day and 12 Months follow-up (both visits taking place in the hospital)

Exclusion Criteria:

1. Patients without signed informed consent / data protection statement (according to requirements of local IRB/IEC)
2. Life expectancy below 12 months
3. Patients with largely incomplete data with respect to the aims of the project
4. Pregnant women at the time of the redo-TAVI

Note: For all patients included a defined core data set will be collected prospectively. All patients being in accordance with above stated inclusion and exclusion criteria and receiving a balloon-expandable transcatheter aortic valve will be included in the extended documentation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an indication for a redo-TAVI procedure considered eligible by the Local Heart Team and the Case Review Board for a SAPIEN family valve implantation.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy: VARC-3 defined device success at 30 days | 30 days
  Determine VARC-3 defined device success at 30 days
  * Technical success
  * Freedom from mortality
  * Freedom from surgery or intervention related to the device or a major vascular or access-related or cardiac structural complication
  * Intended performance of the valve (mean gradient <20 mmHg, peak velocity <3 m/s, Doppler velocity index ≥0.25, and less than moderate aortic regurgitation)
  (Different definitions, in addition to the predefined such as the consideration of higher gradients than 20 mmHg, will be explored)
  These events will be adjudicated. Number and percentage of subjects with device success at 30 days as per VARC-3 definition, along with individual component of the success, will be presented.
Technical success: Technical success (at exit from procedure room) | end of intervention
  Technical success at exit from procedure room defined as:
  * Freedom from mortality
  * Successful access, delivery of the device, and retrieval of the delivery system
  * Correct positioning of a single prosthetic heart valve into the proper anatomical location
  * Freedom from surgery or intervention related to the device (excluding pacemaker) or to a major vascular or access-related, or cardiac structural complication
  Number and percentage of subjects with technical success at exit from procedure room, along with individual component of the success, will be presented.
Safety: VARC-3 defined early safety at 30 days | 30 days
  Determine VARC-3 defined early safety at 30 days:
  * Freedom from all-cause mortality
  * Freedom from all Stroke
  * Freedom from all VARC type 2-4 bleeding
  * Freedom from all major vascular, access-related, or cardiac structural complication
  * Freedom from all acute kidney injury stage III/IV
  * Freedom from all moderate/severe aortic regurgitation
  * Freedom from all new permanent pacemaker implantations due to procedure-related conduction abnormalities
  * Freedom from all surgery/intervention related to the device
  These events will be adjudicated. Number and percentage of subjects with early safety at 30 days as per VARC-3 definition, along with individual component of the success, will be presented.
Procedural Outcomes (30 days) | 30 days
  Procedural outcomes at 30 days, defined as:
  * Clinical and anatomical predictors of technical success (type of SVD [stenosis vs. regurgitation], valve size, implant depth, redo-TAVI balloon dilation, CT and echo-derived variables, etc.)
  * Rate of central and paravalvular regurgitation
  * Valve performance, including residual mean gradient
  * Risk and predictors of coronary obstruction
  Number and percentage of subjects with above specified outcomes at 30 days , along with individual component of the success, will be presented.
Durability of the second aortic THV (30 days) | 30 days
  Determine the durability of the second aortic THV:
  * Subclinical transcatheter heart valve thrombosis at thirty days (when it becomes apparent, but no systematic screening)
  * Endocarditis
  Definition of transcatheter heart valve thrombosis Clinical sequelae of a thromboembolic event (e.g. stroke, TIA, retinal occlusion, other evidence of systemic thromboembolism) or worsening valve stenosis/ regurgitation (e.g. signs of heart failure, syncope) and
  * Haemodynamic valve deterioration Stage 2 or 3 or
  * Confirmatory imaging (CT evidence of HALT† or TEE findings) In the absence of clinical sequelae, both
  * Haemodynamic valve deterioration Stage 3 and
  * Confirmatory imaging (CT evidence of HALT or TEE findings)
  Number and percentage of subjects with above specified criteria at 3 months, along with individual component of the success, will be presented.
Durability of the second aortic THV (3 months) | 3 months
  Determine the durability of the second aortic THV:
  * Subclinical transcatheter heart valve thrombosis at three months (if data obtained, when it becomes apparent, but no systematic screening)
  * Clinical transcatheter heart valve thrombosis at three months (if data obtained)
  * Endocarditis
  For the definition of transcatheter cardiac valve thrombosis, please refer to Outcome 5.
  Number and percentage of subjects with above specified criteria at 3 months, along with individual component of the success, will be presented.
Durability of the second aortic THV (12 months) | 12 months
  Determine the durability of the second aortic THV:
  * Subclinical transcatheter heart valve thrombosis at twelve months (when it becomes apparent, but no systematic screening)
  * Clinical transcatheter heart valve thrombosis at twelve months
  * All-cause mortality, stroke, myocardial infarction, and cardiovascular hospitalization at twelve months
  * Stage II or III structural valve degeneration according to VARC 3 definitions at twelve months (stage I may be documented)
  * Endocarditis
  For the definition of transcatheter cardiac valve thrombosis, please refer to Outcome 5. Number and percentage of subjects with above specified criteria at 12 months , along with individual component of the success, will be presented.
Durability of the second aortic THV (3 years) | 3 years
  Determine the durability of the second aortic THV:
  * Subclinical transcatheter heart valve thrombosis at 3 years (when it becomes apparent, but no systematic screening)
  * Clinical transcatheter heart valve thrombosis at 3 years
  * All-cause mortality, stroke, myocardial infarction, and cardiovascular hospitalization at 3 years
  For the definition of transcatheter cardiac valve thrombosis, please refer to Outcome 5.
Durability of the second aortic THV (5 years) | 5 years
  Determine the durability of the second aortic THV:
  * Subclinical transcatheter heart valve thrombosis at 5 years (when it becomes apparent, but no systematic screening)
  * Clinical transcatheter heart valve thrombosis at 5 years
  * All-cause mortality, stroke, myocardial infarction, and cardiovascular hospitalization at 5 years
  For the definition of transcatheter cardiac valve thrombosis, please refer to Outcome 5.

OTHER OUTCOMES:
Compliance with recommendation | 12 months
  It will be assessed and percentages determined whether participating centers follow the published recommendation (itemized, compliance being voluntary).
Impact of alterations to published recommendations | 12 months
  The impact of potential alterations to the protocol on the procedural outcomes will be elucidated and descriptively described.
Discretionary longer-term follow-up | up to 5 years
  Discretionary longer-term follow-up in terms of durability of the second aortic THV:
  * Subclinical transcatheter heart valve thrombosis
  * Clinically symptomatic transcatheter heart valve thrombosis
  * All-cause mortality, stroke, and cardiovascular hospitalization
  * Stage II or III structural valve degeneration according to VARC 3 definitions
  For the definition of transcatheter cardiac valve thrombosis, please refer to Outcome 5.
  Number and percentage of subjects with above specified criteria with up to 5 years follow-up, along with individual component of the success, will be presented.
Exploratory objectives | 12 months
  Further, not predefined research questions will be explored based on the dataset such as:
  * Hemodynamic outcome of the intervention
  * Applicability of VARC-3 criteria for the redo-TAVI situation
  * Coronary artery obstruction due to valve implantation
  * Coronary artery cannulation (in particular in case of risk plane above ostia)
  * Early and late THV failure predictors (after TAVI and redo-TAVI procedures)
  * CT findings related to THV failure (SVD)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Tarantini, Prof., Principal Investigator — University of Padua Medical School, Padua, Italy; Radoslaw Parma, Dr., Principal Investigator — Medical University of Silesia, Katowice, Poland; Thomas Cuisset, Prof., Study Chair — Centre Hospitalier Universitaire de Timone, Marseille, France; Victoria Delgado, Prof., Study Chair — University Hospital Germans Trias i Pujol, Badalona, Spain; Michael Joner, Prof., Study Chair — German Heart Center, Technical University of Munich, Munich, Germany; Thomas Modine, Prof., Study Chair — Hopital Haut Levêque - Centre Hospitalier Universitaire de Bordeaux, France; Josep Rodés-Cabau, Prof., Study Chair — nstitut Universitaire de Cardiologie et de Pneumologie de Québec, Canada; Francesco Saia, Prof., Study Chair — University Hospital of Bologna, Policlinico S. Orsola-Malpighi, Bologna, Italy; Hector A. Alvarez Covarrubias, MD, Study Chair — Department of Cardiology, Munich Heart Center, Technical University of Munich, Germany; Ginatutas Bieliauskas, MD, Study Chair — Department Interventional Cardiology, The Heart Center, Rigshospitalet, University of Copenhagen, Coppenhagen, Denmark; Luca Nai Fovino, MD, Study Chair — Department of Cardiac, Thoracic, Vascular Sciences and Public Health, University of Padua Medical School, Padua, Italy; Eric Van Belle, MD, Study Chair — Interventional Cardiology, Centre Hospitalier Universitaire de Lille, France; Rafał Wolny, MD, Study Chair — Department of Interventional Cardiology and Angiology, National Institute of Cardiology, Warsaw, Poland
Locations (62):
- Austria (4):
  - LKH-University Hospital and Medical University of Graz, Graz
  - Kepler University Clinic Linz, Linz
  - University Hospital St. Pölten, Sankt Pölten
  - Medical University of Vienna, Vienna
- Canada (3):
  - McGill University Health Centre, Montreal
  - Institut Universitaire de Cardiologie et de Pneumologie, Québec
  - St. Paul's Hospital, Vancouver, Vancouver
- France (13):
  - Centre Hospitalier Universitaire de Bordeaux, Bordeaux
  - Centre Hospitalier Universitaire de Clermont-Ferrand, Clermont-Ferrand
  - Centre Hospitalier Universitaire de Lille, Lille
  - Hospices Civils de Lyon, Lyon
  - Hôpitaux Universitaires de Marseille Timone, Marseille
  - Jacques Cartier Private Hospital, Massy, Massy
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - Hôpital Européen Georges-Pompidou, Paris
  - Hôpital Bichat-Claude-Bernard, Paris
  - Centre hospitalier universitaire de Rennes, Rennes
  - Centre Hospitalier Universitaire de Rouen, Roubaix
  - Clinique de la Porte de Paris (CCN), Saint-Denis
  - Centre Hospitalier Universitaire de Toulouse, Toulouse
- Germany (10):
  - University Heart Center Freiburg Bad Krozingen, Bad Krozingen
  - Kerckhoff-Klinik GmbH, UKGM GmbH, Bad Nauheim
  - Heart and Diabetes Center North Rhine-Westphalia, Bad Oeynhausen
  - German Heart Center of Charité Berlin, Berlin
  - BG University Hospital Bergmannsheil gGmbH, Bochum
  - University Hospital of Duesseldorf, Düsseldorf
  - Elisabeth Hospital, Essen, Essen
  - German Heart Centre Munich, Munich
  - Robert-Bosch-Hospital, Stuttgart, Stuttgart
  - University Hospital Ulm, Ulm
- Tel Aviv Medical Center, Tel Aviv, Israel
- Italy (11):
  - AOU Ospedali Riuniti Ancona, Umberto I, G. M. Lancisi, G. Salesi, Ancona
  - IRCCS Azienda Ospedaliero Universitaria di Bologna, Bologna
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia, Brescia
  - Careggi Hospital, Florence
  - IRCCS Ospedale Galeazzi Sant'Ambrogio, Milan
  - Azienda Ospedale-Università Padova (AOUP), Padua
  - Azienda Ospedaliero-Universitaria Pisana, Pisa
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - Policlinici universitari | Sapienza Università di Roma, Roma
  - Università degli Studi di Trieste, Trieste
  - Ospedale San Bortolo di Vicenza, Vicenza
- St. Antonius Ziekenhuis, Nieuwegein, Nieuwegein, Netherlands
- Poland (7):
  - Medical University of Bialystok, Bialystok
  - University Clinical Centre of Gdańsk, Gdansk
  - Medical University of Silesia, Katowice
  - University Hospital of Kraków, Krakow
  - Medical University of Warsaw, Warsaw
  - Institute of Cardiology Warsaw, Warsaw
  - Wroclaw Medical University, Wroclaw
- Portugal (2):
  - Hospital de Santa Cruz, Carnaxide-Lisabon, Carnaxide
  - Centro Hospitalar Vila Nova de Gaia / Espinho, Vila Nova de Gaia
- Spain (7):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital University Germans Trias i Pujol, Barcelona
  - Hospital Universitario de León, León
  - Hospital Clinico Universitario San Carlos, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Álvaro Cunqueiro, Vigo, Vigo
- Switzerland (3):
  - University Hospital of Basel, Basel
  - Hôpitaux universitaires de Genève, Geneva
  - Centre hospitalier universitaire vaudois et Université de Lausanne, Lausanne

IPD SHARING:
Plan to Share IPD: No
no individual participant data (IPD) will be shared

REFERENCES:
- [Background] VARC-3 WRITING COMMITTEE; Genereux P, Piazza N, Alu MC, Nazif T, Hahn RT, Pibarot P, Bax JJ, Leipsic JA, Blanke P, Blackstone EH, Finn MT, Kapadia S, Linke A, Mack MJ, Makkar R, Mehran R, Popma JJ, Reardon M, Rodes-Cabau J, Van Mieghem NM, Webb JG, Cohen DJ, Leon MB. Valve Academic Research Consortium 3: updated endpoint definitions for aortic valve clinical research. Eur Heart J. 2021 May 14;42(19):1825-1857. doi: 10.1093/eurheartj/ehaa799. PMID 33871579
- [Background] Tarantini G, Delgado V, de Backer O, Sathananthan J, Treede H, Saia F, Blackman D, Parma R. Redo-Transcatheter Aortic Valve Implantation Using the SAPIEN 3/Ultra Transcatheter Heart Valves-Expert Consensus on Procedural Planning and Techniques. Am J Cardiol. 2023 Apr 1;192:228-244. doi: 10.1016/j.amjcard.2023.01.010. Epub 2023 Jan 27. PMID 36710143
- [Background] Leon MB, Smith CR, Mack M, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Brown DL, Block PC, Guyton RA, Pichard AD, Bavaria JE, Herrmann HC, Douglas PS, Petersen JL, Akin JJ, Anderson WN, Wang D, Pocock S; PARTNER Trial Investigators. Transcatheter aortic-valve implantation for aortic stenosis in patients who cannot undergo surgery. N Engl J Med. 2010 Oct 21;363(17):1597-607. doi: 10.1056/NEJMoa1008232. Epub 2010 Sep 22. PMID 20961243
- [Background] Smith CR, Leon MB, Mack MJ, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Williams M, Dewey T, Kapadia S, Babaliaros V, Thourani VH, Corso P, Pichard AD, Bavaria JE, Herrmann HC, Akin JJ, Anderson WN, Wang D, Pocock SJ; PARTNER Trial Investigators. Transcatheter versus surgical aortic-valve replacement in high-risk patients. N Engl J Med. 2011 Jun 9;364(23):2187-98. doi: 10.1056/NEJMoa1103510. Epub 2011 Jun 5. PMID 21639811
- [Background] Toggweiler S, Wood DA, Rodes-Cabau J, Kapadia S, Willson AB, Ye J, Cheung A, Leipsic J, Binder RK, Gurvitch R, Freeman M, Thompson CR, Svensson LG, Dumont E, Tuzcu EM, Webb JG. Transcatheter valve-in-valve implantation for failed balloon-expandable transcatheter aortic valves. JACC Cardiovasc Interv. 2012 May;5(5):571-577. doi: 10.1016/j.jcin.2012.03.008. PMID 22625197
- [Background] Kamioka N, Caughron H, Corrigan F, Block P, Babaliaros V. Supra-annular valve strategy for an early degenerated transcatheter balloon-expandable heart valve. Catheter Cardiovasc Interv. 2018 Dec 1;92(7):1458-1460. doi: 10.1002/ccd.27506. Epub 2018 Jan 23. PMID 29359409
- [Background] Webb JG, Mack MJ, White JM, Dvir D, Blanke P, Herrmann HC, Leipsic J, Kodali SK, Makkar R, Miller DC, Pibarot P, Pichard A, Satler LF, Svensson L, Alu MC, Suri RM, Leon MB. Transcatheter Aortic Valve Implantation Within Degenerated Aortic Surgical Bioprostheses: PARTNER 2 Valve-in-Valve Registry. J Am Coll Cardiol. 2017 May 9;69(18):2253-2262. doi: 10.1016/j.jacc.2017.02.057. PMID 28473128
- [Background] Deeb GM, Chetcuti SJ, Reardon MJ, Patel HJ, Grossman PM, Schreiber T, Forrest JK, Bajwa TK, O'Hair DP, Petrossian G, Robinson N, Katz S, Hartman A, Dauerman HL, Schmoker J, Khabbaz K, Watson DR, Yakubov SJ, Oh JK, Li S, Kleiman NS, Adams DH, Popma JJ. 1-Year Results in Patients Undergoing Transcatheter Aortic Valve Replacement With Failed Surgical Bioprostheses. JACC Cardiovasc Interv. 2017 May 22;10(10):1034-1044. doi: 10.1016/j.jcin.2017.03.018. PMID 28521921
- [Background] Kopp-Schneider A, Wiesenfarth M, Witt R, Edelmann D, Witt O, Abel U. Monitoring futility and efficacy in phase II trials with Bayesian posterior distributions-A calibration approach. Biom J. 2019 May;61(3):488-502. doi: 10.1002/bimj.201700209. Epub 2018 Sep 2. PMID 30175405
- See also: The ReTAVi Registry webpage provides you with general details about the trial and gives you an overview of participating trial sites. — https://www.retavi-registry.com/